CLINICAL TRIAL: NCT05617118
Title: Evaluation of Efficacy and Safety of Oral Baclofen Taking in Comparison With Botulinum Toxin A Injections in Myofascial Pelvic Pain Syndrome. Prospective Multicenter Cohort Study.
Brief Title: BTA vs Baclofen for Pelvic Myofascial Pain Syndrome
Acronym: BvsB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saint Petersburg State University, Russia (Other)
Collaborators: Ural State Medical University (Other)
Responsible Party: Principal Investigator, Gleb Kovalev, Kovalev Gleb, head of outpatient urology department, urologist, Saint Petersburg State University, Russia
Other Study IDs: 22/30 301
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Chronic Pain; Chronic Pelvic Pain Syndrome; Myofascial Pain Syndrome; Myofascial Trigger Point Pain; Pelvic Floor Disorders
MeSH Terms: conditions — Chronic Pain; Myofascial Pain Syndromes; Pelvic Floor Disorders | interventions — Baclofen; Botulinum Toxins, Type A; incobotulinumtoxinA; abobotulinumtoxinA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baclofen: A cohort of patients who have not previously received baclofen will be offered a course of the drug therapy at a dosage of 10 mg according to the scheme:
  1-3 days - 1 tablet per day; 4-6 days - 2 tablets per day; 7-9 days - 3 tablets per day; 10 days and then 4 tablets per day (morning and evening).
  Interventions: Drug: Baclofen 10mg
- BTA: A cohort of patients who previously received baclofen and canceled the course due to the development of side effects and/or individual intolerance, or who have contraindications to the use of this drug, will receive several injections with a total volume of 100 units. botulinum toxin type "A" in dilution up to 20 ml, distributed at the trigger points of the pelvic floor muscles.
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Baclofen 10mg — Baclofen is a medication, a central myorelaxant, a GABAb stimulator.
  Other Names: Baclosan
  Groups: Baclofen
Drug: Botulinum toxin type A — Botulinum toxin, often shortened to BoNT, is a neurotoxic protein produced by the bacterium Clostridium botulinum and related species.
  Other Names: Botox, Xeomin, Dysport
  Groups: BTA

SUMMARY:
The aim of the study is to test the hypothesis that oral taking of baclofen in therapeutic dosage for 60 days is equally effective as injection of botulinum toxin type "A" in the area of trigger points of the pelvic muscles.

DETAILED DESCRIPTION:
Chronic pelvic pain syndrome (CPPS) is an extremely common disease. The exact epidemiology and socio-economic impact cannot be determined due to its heterogeneity. Thus, according to population studies, CPPS can occur in 12.4% of women aged 18-50 years [1]. In turn, myofascial pelvic pain syndrome (MPPS) is often an underappreciated and untreated component of CPPS that occurs in at least 23% of patients and causes their complaints [2]. In men diagnosed with chronic prostatitis, in 92% of cases, complaints are caused by muscle spasm and pain in muscle structures, mistakenly interpreted by the patient as prostate pain [3]. Often, myofascial syndrome is idiopathic and is associated with problems in the musculoskeletal system. However, in some cases, the primary source is a urological, gynecological or proctological disease. The syndrome is characterized by the appearance of trigger points (TP) - "nodules" in the thickness of striated muscles, which cause distinct local soreness during palpation [4].

Treatment of this condition is complex: it includes training in relaxation of the pelvic muscles using a biofeedback therapy [5], myofascial release [6] and drug therapy. One of the drugs actively used in neurology is baclofen [7]. This drug reduces the spasticity of striated muscles. Despite the widespread using of baclofen in the treatment of neurological conditions accompanied by increased muscle tone, there are no qualitative studies evaluating its effectiveness in chronic pelvic pain syndrome.

If conservative therapy is ineffective, injections of botulinum toxin type "A" (BTA) into TP on pelvic floor muscles are the method of choice [8]. This method is a third-line treatment: thus, according to the meta-analysis of Fang Yuan Luo et al., which includes 5 RCTs and 12 observational studies, there is not enough convincing data for using BTA as the first line of treatment [9]. At the same time, there are a number of studies in which the effect of the introduction of BTA was comparable to the introduction of local anesthetics [10] and saline solution [11].

Thus, despite the inconsistency of the methods, a comparative study of the efficacy and safety of these drugs, as well as the quality of life of patients after treatment, is of interest.

ELIGIBILITY:
Inclusion Criteria:

* Myofascial pain syndrome (presence of trigger points), confirmed by palpation during examination.
* Ineffectiveness (with subsequent discontinuation) of at least one treatment method, including outpatient physiotherapy and /or oral analgesics, or NSAIDs.

Exclusion Criteria:

* The presence of any organic disease of the pelvic organs requiring active treatment, confirmed by anamnesis, consultation of a specialist (urologist, proctologist, gynecologist) and one of the objective imaging methods: CT, MRI, endoscopical or laboratory methods: general urine analysis or prostate secretion analysis. Such diseases include interstitial cystitis / SBMP, chronic prostatitis types I, II, IIIA according to the NIH classification.
* The presence in the anamnesis of the fact of previously conducted therapy with baclofen or injection of botulinum toxin type "A" into the pelvic floor muscles.
* Individual intolerance to botulinum toxin type "A" and /or baclofen.
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with long-term chronic pelvic pain syndrome who have not previously received targeted treatment for myofascial pelvic pain syndrome
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
PGI-I | 60 days
  Patients Global Impression of Improvement (PGI-I). The PGI-I is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1. Very much better to 7. Very much worse.

SECONDARY OUTCOMES:
VAS | 14, 30, 60 days
  Visual Analogue Scale (VAS). The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best). The line is divided into 10 sections. 1 section = 1 point. The more points, the more pronounced the pain syndrome - the worse outcome
The Lamont Scale | 14, 30, 60 days
  The Lamont scale was developed to aide in the diagnosis of vaginismus. The five degrees of severity are defined. The more points, the more pronounced the patient's reaction to the examination in the gynecological chair. Points from 1 to 5. The The higher the score, the more pronounced the vaginismus and fear of examination. Minimum score = 0. Maximum score = 5. The lower score, the better outcome
IPSS/QoL | 14, 30, 60 days
  International Prostate Symptom Score (IPSS). The IPSS questionnaire evaluates the impact of lower urinary tract symptoms on the patient's quality of life. It consists of 8 questions. Questionts evaluates whether the patient has symptoms of incomplete emptying of the bladder and ranges from 0 to 5 points. The increase in scores is directly proportional to the increase in symptoms. Minimum score = 0. Maximum score = 41. The lower score, the better outcome
Clavien-Dindo Complication rate | 14, 30, 60 days
  The development of complications from therapy that require its termination

CONTACTS AND LOCATIONS:
Locations (1):
- SBPSU, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available upon request after the study is completed

REFERENCES:
- [Background] Zondervan K, Barlow DH. Epidemiology of chronic pelvic pain. Baillieres Best Pract Res Clin Obstet Gynaecol. 2000 Jun;14(3):403-14. doi: 10.1053/beog.1999.0083. PMID 10962634
- [Background] Tu FF, As-Sanie S, Steege JF. Prevalence of pelvic musculoskeletal disorders in a female chronic pelvic pain clinic. J Reprod Med. 2006 Mar;51(3):185-9. PMID 16674013
- [Background] Zermann D, Ishigooka M, Doggweiler R, Schmidt R. Chronic prostatitis: A myofascial pain syndrome? Infections in Urology 1999;12:84-92
- [Background] Jha S, Toozs-Hobson P, Roper JC, Gurung S, Brair A, Bach F. Botulinum injections for myofascial pelvic pain. Int Urogynecol J. 2021 May;32(5):1151-1156. doi: 10.1007/s00192-020-04435-w. Epub 2020 Jul 21. PMID 32696187
- [Background] Hite M, Curran T. Biofeedback for Pelvic Floor Disorders. Clin Colon Rectal Surg. 2021 Jan;34(1):56-61. doi: 10.1055/s-0040-1714287. Epub 2020 Sep 4. PMID 33536850
- [Background] Peñas CF de las, Campo MS, Carnero JF, Page JCM. Manual therapies in myofascial trigger point treatment: A systematic review. Journal of Bodywork and Movement Therapies 2005;9:27-34. doi:10.1016/j.jbmt.2003.11.001.
- [Background] Chang WJ. Muscle Relaxants for Acute and Chronic Pain. Phys Med Rehabil Clin N Am. 2020 May;31(2):245-254. doi: 10.1016/j.pmr.2020.01.005. Epub 2020 Mar 13. PMID 32279727
- [Background] Morrissey D, El-Khawand D, Ginzburg N, Wehbe S, O'Hare P 3rd, Whitmore K. Botulinum Toxin A Injections Into Pelvic Floor Muscles Under Electromyographic Guidance for Women With Refractory High-Tone Pelvic Floor Dysfunction: A 6-Month Prospective Pilot Study. Female Pelvic Med Reconstr Surg. 2015 Sep-Oct;21(5):277-82. doi: 10.1097/SPV.0000000000000177. PMID 25900057
- [Background] Luo FY, Nasr-Esfahani M, Jarrell J, Robert M. Botulinum toxin injection for chronic pelvic pain: A systematic review. Acta Obstet Gynecol Scand. 2020 Dec;99(12):1595-1602. doi: 10.1111/aogs.13946. Epub 2020 Jul 16. PMID 32597494
- [Background] Levesque A, Ploteau S, Michel F, Siproudhis L, Bautrant E, Eggermont J, Rabischong B, Volteau C, Perrouin-Verbe MA, Labat JJ. Botulinum toxin infiltrations versus local anaesthetic infiltrations in pelvic floor myofascial pain: Multicentre, randomized, double-blind study. Ann Phys Rehabil Med. 2021 Jan;64(1):101354. doi: 10.1016/j.rehab.2019.12.009. Epub 2020 Jan 22. PMID 31981833
- [Background] Parsons BA, Goonewardene S, Dabestani S, Pacheco-Figueiredo L, Yuan Y, Zumstein V, Cottrell AM, Borovicka J, Dinis-Oliveira P, Berghmans B, Elneil S, Hughes J, Messelink BEJ, de C Williams AC, Baranowski AP, Engeler DS. The Benefits and Harms of Botulinum Toxin-A in the Treatment of Chronic Pelvic Pain Syndromes: A Systematic Review by the European Association of Urology Chronic Pelvic Pain Panel. Eur Urol Focus. 2022 Jan;8(1):320-338. doi: 10.1016/j.euf.2021.01.005. Epub 2021 Jan 30. PMID 33526405
- [Background] Cook D, Lauzier F, Rocha MG, Sayles MJ, Finfer S. Serious adverse events in academic critical care research. CMAJ. 2008 Apr 22;178(9):1181-4. doi: 10.1503/cmaj.071366. No abstract available. PMID 18427095